CLINICAL TRIAL: NCT02598492
Title: Imputation of PaO2 From SaO2 in the Respiratory Component of the Sequential Organ Failure Assessment (SOFA) Score
Brief Title: Imputation of PaO2 From SaO2
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Guangzhou Red Cross Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peter Chuanyi Hou, Associate Physician, Brigham and Women's Hospital
Other Study IDs: 2015P001945
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Failure
Keywords: Mechanical Ventilator
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imputation of SF to PF: Patients required invasive mechanical ventilation within 6 hours after intubation
  Interventions: Other: arterial blood gas

INTERVENTIONS:
Other: arterial blood gas — Just record clinical lab data
  Other Names: oxygena saturation

SUMMARY:
The aims of this study are (1) to find out the relationship between PaO2 and SaO2 among mechanically ventilated patients and (2) to create a reliable system to utilize SF ratios to impute the PF ratios in assessing the respiratory parameter of the SOFA score.

DETAILED DESCRIPTION:
The Sequential Organ Failure Assessment (SOFA) score is validated as a measure of severity of illness over time in intensive care unit (ICU) patients and can be used to follow the course of organ dysfunction and response to treatment1. SOFA has become a frequently used scoring system of patients in multi-organ failure, given its high sensitivity and specificity as a predictor of morbidity and mortality in critically ill patients2. The severity of respiratory dysfunction is measured in the SOFA score by PaO2/FiO2 (PF) ratio, which is also used as a measure of severity of hypoxemia in patients with acute respiratory distress syndrome (ARDS).

An invasive sampling of arterial blood gas (ABG) is required to measure the PaO2 for the PF. Often, patients with less severe hypoxemia may not clinically undergo ABG testing on a routine basis; hence the clinical and research utility of the SOFA scoring system is reduced. Furthermore, previous studies revealed concerns about anemia following repeated blood sampling; hence, the tendency to implement less invasive approaches have led to less frequent ABG measurements in critically ill patients3. However, almost all ICU patients are monitored with pulse oximeters, which measure the percent saturation of hemoglobin with oxygen (SpO2). Whether SpO2 can be used to impute PaO2 for determining the PF ratio has not been robustly evaluated in a prospective study of critically ill patients.

Prior work investigating the association between PaO2 and SpO2 includes a post hoc study of ARDS Network patients4. This study excluded patients at altitude, used a linear model for a highly non-linear relationship, and could not determine whether SpO2 and PaO2 were simultaneously measured. A similar approach was applied to ARDS Network patients to derive an SpO2-based respiratory subscore of the SOFA score5. Several similar, retrospective studies have been performed in mechanically ventilated children, consistently using linear models of correlation between SF and PF ratios, with similar limitations6-9.

The Ellis inversion10 of the Severinghaus equation11 provides a useful non-linear method for imputing PaO2 from SaO2. This technique has been used in multiple cohorts of patients with pneumonia12-14. This simple calculation can be improved by incorporating PaCO2 and pH values, which could be available from venous blood gases that may be obtained in patients without arterial catheters. Because Severinghaus/Ellis estimates SaO2, a method for estimating SaO2 from SpO2 is necessary. There is no current validated and reliable method for calculating SaO2 on the basis of a measured SpO2. Skin pigmentation affects accuracy of SpO2, as do sex and oximeter type15,16.

The aims of this study are (1) to find out the relationship between PaO2 and SaO2 among mechanically ventilated patients and (2) to create a reliable system to utilize SF ratios to impute the PF ratios in assessing the respiratory parameter of the SOFA score.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated patient in a participating ICU or ED.
2. Arterial blood gas ordered and obtained for clinical reasons.

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults > 18 years old who are invasively mechanically ventilated in an ED or ICU
Sampling Method: Non-Probability Sample
Enrollment: 646 (Actual)
Dates: Start 2015-09-01; Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between PaO2 and SaO2 among mechanically ventilated patients | one year

SECONDARY OUTCOMES:
To utilize SF ratios to impute the PF ratios in assessing the respiratory parameter of the SOFA score | one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Hou, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- China (2):
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - PLA General Hospital, Beijing

REFERENCES:
- [Result] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Result] Vincent JL, Ferreira F, Moreno R. Scoring systems for assessing organ dysfunction and survival. Crit Care Clin. 2000 Apr;16(2):353-66. doi: 10.1016/s0749-0704(05)70114-7. PMID 10768086
- [Result] Ferguson ND, Frutos-Vivar F, Esteban A, Fernandez-Segoviano P, Aramburu JA, Najera L, Stewart TE. Acute respiratory distress syndrome: underrecognition by clinicians and diagnostic accuracy of three clinical definitions. Crit Care Med. 2005 Oct;33(10):2228-34. doi: 10.1097/01.ccm.0000181529.08630.49. PMID 16215375
- [Result] Rice TW, Wheeler AP, Bernard GR, Hayden DL, Schoenfeld DA, Ware LB; National Institutes of Health, National Heart, Lung, and Blood Institute ARDS Network. Comparison of the SpO2/FIO2 ratio and the PaO2/FIO2 ratio in patients with acute lung injury or ARDS. Chest. 2007 Aug;132(2):410-7. doi: 10.1378/chest.07-0617. Epub 2007 Jun 15. PMID 17573487
- [Result] Pandharipande PP, Shintani AK, Hagerman HE, St Jacques PJ, Rice TW, Sanders NW, Ware LB, Bernard GR, Ely EW. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. Crit Care Med. 2009 Apr;37(4):1317-21. doi: 10.1097/CCM.0b013e31819cefa9. PMID 19242333
- [Result] Khemani RG, Patel NR, Bart RD 3rd, Newth CJL. Comparison of the pulse oximetric saturation/fraction of inspired oxygen ratio and the PaO2/fraction of inspired oxygen ratio in children. Chest. 2009 Mar;135(3):662-668. doi: 10.1378/chest.08-2239. Epub 2008 Nov 24. PMID 19029434
- [Result] Khemani RG, Thomas NJ, Venkatachalam V, Scimeme JP, Berutti T, Schneider JB, Ross PA, Willson DF, Hall MW, Newth CJ; Pediatric Acute Lung Injury and Sepsis Network Investigators (PALISI). Comparison of SpO2 to PaO2 based markers of lung disease severity for children with acute lung injury. Crit Care Med. 2012 Apr;40(4):1309-16. doi: 10.1097/CCM.0b013e31823bc61b. PMID 22202709
- [Result] Thomas NJ, Shaffer ML, Willson DF, Shih MC, Curley MA. Defining acute lung disease in children with the oxygenation saturation index. Pediatr Crit Care Med. 2010 Jan;11(1):12-7. doi: 10.1097/PCC.0b013e3181b0653d. PMID 19561556
- [Result] Lobete C, Medina A, Rey C, Mayordomo-Colunga J, Concha A, Menendez S. Correlation of oxygen saturation as measured by pulse oximetry/fraction of inspired oxygen ratio with Pao2/fraction of inspired oxygen ratio in a heterogeneous sample of critically ill children. J Crit Care. 2013 Aug;28(4):538.e1-7. doi: 10.1016/j.jcrc.2012.12.006. Epub 2013 Feb 8. PMID 23395312
- [Result] Ellis RK. Determination of PO2 from saturation. J Appl Physiol (1985). 1989 Aug;67(2):902. doi: 10.1152/jappl.1989.67.2.902. No abstract available. PMID 2793692
- [Result] Severinghaus JW. Simple, accurate equations for human blood O2 dissociation computations. J Appl Physiol Respir Environ Exerc Physiol. 1979 Mar;46(3):599-602. doi: 10.1152/jappl.1979.46.3.599. PMID 35496
- [Result] Lanspa MJ, Jones BE, Brown SM, Dean NC. Mortality, morbidity, and disease severity of patients with aspiration pneumonia. J Hosp Med. 2013 Feb;8(2):83-90. doi: 10.1002/jhm.1996. Epub 2012 Nov 26. PMID 23184866
- [Result] Dean NC, Jones JP, Aronsky D, Brown S, Vines CG, Jones BE, Allen T. Hospital admission decision for patients with community-acquired pneumonia: variability among physicians in an emergency department. Ann Emerg Med. 2012 Jan;59(1):35-41. doi: 10.1016/j.annemergmed.2011.07.032. Epub 2011 Sep 9. PMID 21907451
- [Result] Brown SM, Jones BE, Jephson AR, Dean NC; Infectious Disease Society of America/American Thoracic Society 2007. Validation of the Infectious Disease Society of America/American Thoracic Society 2007 guidelines for severe community-acquired pneumonia. Crit Care Med. 2009 Dec;37(12):3010-6. doi: 10.1097/CCM.0b013e3181b030d9. PMID 19789456
- [Result] Bickler PE, Feiner JR, Severinghaus JW. Effects of skin pigmentation on pulse oximeter accuracy at low saturation. Anesthesiology. 2005 Apr;102(4):715-9. doi: 10.1097/00000542-200504000-00004. PMID 15791098
- [Result] Feiner JR, Severinghaus JW, Bickler PE. Dark skin decreases the accuracy of pulse oximeters at low oxygen saturation: the effects of oximeter probe type and gender. Anesth Analg. 2007 Dec;105(6 Suppl):S18-S23. doi: 10.1213/01.ane.0000285988.35174.d9. PMID 18048893
- [Result] Utada K, Matayoshi Y, Fujita F, Nakamura K, Matsuda N, Kondoh K, Tamura H. [Equilibration period for PaO2 following alteration of FIO2 in mechanically ventilated patients]. Masui. 2000 Mar;49(3):312-5. Japanese. PMID 10752330
- [Result] Fildissis G, Katostaras T, Moles A, Katsaros A, Myrianthefs P, Brokalaki H, Tsoumakas K, Baltopoulos G. Oxygenation equilibration time after alteration of inspired oxygen in critically ill patients. Heart Lung. 2010 Mar-Apr;39(2):147-52. doi: 10.1016/j.hrtlng.2009.06.009. Epub 2009 Aug 13. PMID 20207275